CLINICAL TRIAL: NCT00023387
Title: Intensive Pharmacokinetic Study of Three Doses of Rifapentine (600, 900 and 1200mg) During Continuation Phase Therapy of Tuberculosis in HIV-Negative Adults
Brief Title: TBTC Study 25PK: Intensive Pharmacokinetic Study of Three Doses of Rifapentine and 25-Desacetyl Rifapentine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDC-NCHSTP-2558; TBTC Study 25PK
Record Dates: First submitted 2001-09-06; First posted 2001-09-10 (Estimated); Last update posted 2005-09-13 (Estimated); Status verified 2005-09

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — rifapentine; 25-desacetylrifapentine; Isoniazid

INTERVENTIONS:
Drug: Rifapentine
Drug: 25-desacetyl Rifapentine
Drug: Isoniazid

SUMMARY:
Primary objective: To compare the pharmacokinetics of rifapentine and 25-desacetyl rifapentine at three different doses: 600 mg, 900 mg, and 1200 mg.

Secondary objective: To describe any correlation between pharmacokinetic parameters of three different doses of rifapentine plus a standard dose of isoniazid and the occurrence of toxicity attributed to anti-tuberculosis treatment.

DETAILED DESCRIPTION:
We will enroll 24-36 patients, 8-12 at each dose of 600, 900 and 1200 mg rifapentine Admissions for pharmacokinetic studies will take place during the continuation phase of tuberculosis therapy. Patients participating in a double-blinded trial of the tolerability and safety of higher doses of rifapentine during continuation phase therapy and consenting to participate in the pharmacokinetic study may be admitted to a Clinical Research Center (CRC) to allow for frequent blood sampling over a 24-hour period. Otherwise, patients will be evaluated in the clinic.

ELIGIBILITY:
Inclusion:

Patients enrolled in TBTC Study 25 Informed consent

Exclusion:

Severe anemia (Hct <25%) Any severe adverse event related to study drugs in TBTC Study 25

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2000-03; Study Completion 2001-05

PRIMARY OUTCOMES:
Compare the pharmacokinetics of rifapentine and 25-desacetyl rifapentine at three difference doses: 600 mg, 900 mg, and 1200 mg

SECONDARY OUTCOMES:
Describe any correlation between pharmacokinetic parameters of three different doses of rifapentine plus a standard dose of isoniazid and the occurrence of toxicity attributed to anti-tuberculosis treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Weiner, MD, Principal Investigator — Audie L. Murphy VA Medical Center, San Antonio TX
Locations (23):
- United States (20):
  - Central Arkansas Veterans Health System, Little Rock, Arkansas
  - LA County/USC Medical Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Denver Department of Public Health and Hospitals, Denver, Colorado
  - Washington, D.C. VAMC, Washington D.C., District of Columbia
  - Chicago VA Medical Center (Lakeside), Chicago, Illinois
  - Hines VA Medical Center, Hines, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - New Jersey Medical School, Newark, New Jersey
  - New York University School of Medicine, New York, New York
  - Columbia University/Presbyterian Medical Center, New York, New York
  - Harlem Hospital Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Nashville VA Medical Center, Nashville, Tennessee
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Thomas Street Clinic, Houston, Texas
  - Audi L. Murphy VA Hospital, San Antonio, Texas
  - Seattle King County Health Department, Seattle, Washington
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Montreal Chest Institute McGill University, Montreal, Quebec

REFERENCES:
- [Background] Weiner M, Bock N, Peloquin CA, Burman WJ, Khan A, Vernon A, Zhao Z, Weis S, Sterling TR, Hayden K, Goldberg S; Tuberculosis Trials Consortium. Pharmacokinetics of rifapentine at 600, 900, and 1,200 mg during once-weekly tuberculosis therapy. Am J Respir Crit Care Med. 2004 Jun 1;169(11):1191-7. doi: 10.1164/rccm.200311-1612OC. Epub 2004 Feb 12. PMID 14962821
- See also: (Click here for more information about the Tuberculosis Trials Consortium(TBTC) — http://www.cdc.gov/nchstp/tb/tbtc/